CLINICAL TRIAL: NCT00795600
Title: A Multi-centre, Open-labelled, Randomised, Two-group Parallel Trial Comparing the Change in Fat Distribution in Overweight and Obese Subjects With Type 2 Diabetes After 26 Weeks of Treatment With Insulin Detemir Once Daily Versus Insulin NPH Once Daily, Both With Insulin Aspart at Mealtimes
Brief Title: Comparison of the Change in Fat Distribution in Overweight and Obese Subjects With Type 2 Diabetes After Insulin Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-3614; 2008-003739-19 (EudraCT Number)
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Results first posted 2013-06-17 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin detemir (Experimental): Insulin detemir injected subcutaneously (s.c.) in the evening in combination with insulin aspart injected s.c. as mealtime insulin for 26 weeks
  Interventions: Drug: insulin detemir
- insulin NPH (Active Comparator): Insulin isophane (Neutral Protamine Hagedorn, NPH) injected subcutaneously (s.c.) in the evening in combination with insulin aspart injected s.c. as mealtime insulin for 26 weeks
  Interventions: Drug: insulin NPH

INTERVENTIONS:
Drug: insulin detemir — Insulin detemir once daily plus insulin aspart at mealtime
  Arms: insulin detemir
Drug: insulin NPH — Insulin NPH once daily plus insulin aspart at mealtime
  Arms: insulin NPH

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to compare the change in trunk fat mass, assessed by Double Energy X-ray Absorptiometry (DEXA) after 26 weeks of treatment with insulin detemir or insulin NPH (Neutral Protamine Hagedorn) (both combined with insulin aspart at the main meals) in overweight and obese subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes who have been treated with 2 or 3 doses of insulin (one of them must be a premix) for at least 3 months prior to inclusion in trial
* Glycosylated haemoglobin (HbA1c) between 7.0-11.0 %
* Body Mass Index (BMI) between 27.5-40 kg/m^2

Exclusion Criteria:

* Treatment with any oral antidiabetic drugs (OADs) in the last 6 months except metformin (subjects currently treated with metformin within the interval of 1000 - 2550 mg daily may be included in the trial. The dose should have remained unchanged for a period of 2 months prior to randomisation and should be expected to remain unchanged throughout the trial period)
* Use of approved weight lowering pharmacotherapy (e.g. orlistat, sibutramin, rimonabant) or obesity induced by drug treatment (e.g. corticosteroids, Non-steroidal anti-inflammatory drugs (NSAIDs), tricyclic anti-depressants, atypical anti-psychotics)
* Previous or planned surgical treatment of obesity
* Total daily insulin dose higher or equal 2 IU/kg
* Proliferative retinopathy or maculopathy that has required acute treatment within the last six months
* Receipt of any investigational drug within 1 month prior to this trial
* Cardiac disease defined according to New York Heart Association (NYHA) class III or IV, unstable angina pectoris and/or myocardial infarction within the last 6 months previous to the selection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Málaga, Spain

REFERENCES:
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from 29-Apr-2009 until 02-Feb-2010. 5 sites in Spain.
Period: Overall Study
Arm/Group | Insulin Detemir | Insulin NPH
Started | 25 | 35
Exposed to Drug | 24 (1 patient did not take study medication because the patient withdrew consent) | 35
Completed | 21 | 31
Not Completed | 4 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Unclassified | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Detemir | Insulin NPH | Total
Number analyzed (Participants) | 24 | 35 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 6 | 17 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.63 (8.87) | 63.74 (9.39) | 62.47 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 19 | 30
  Male | 13 | 16 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 24 | 35 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 35 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 24 | 35 | 59
Duration of diabetes [Mean (Standard Deviation); unit: years] — Number of years since diagnosis
  years | 13.58 (6.68) | 17.43 (9.00) | 15.86 (8.29)
Diabetic complication at baseline, nephropathy (common risk factor in uncontrolled diabetes) [Number; unit: participants]
  Yes | 4 | 5 | 9
  No | 20 | 30 | 50
Diabetic complication at baseline, neuropathy (common risk factor in uncontrolled diabetes) [Number; unit: participants]
  Yes | 5 | 7 | 12
  No | 19 | 28 | 47
Diabetic complication at baseline, retinopathy (common risk factor in uncontrolled diabetes) [Number; unit: participants]
  Yes | 11 | 16 | 27
  No | 13 | 19 | 32
Diabetic complication at baseline, macroangiopathy [Number; unit: participants]
  Yes | 4 | 12 | 16
  No | 20 | 23 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Trunk Fat Mass (Defined as Peripheral Fat Ratio)
Description: Percentage of change of trunk fat mass as the dependent variable, baseline value (trunk fat mass at week 0) as covariate, treatment with metformin (yes/no) and gender (male/female) as effect and the treatment received (insulin detemir/insulin NPH) as the main factor.
Time Frame: week 0, week 26
Population: Intention-To-Treat (ITT) analysis set using LOCF (Last Observation Carried Forward) is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in the change in trunk fat mass at week 26.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
percent change | 0.366 (2.785) | 1.011 (2.158)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; The primary objective and endpoint of the trial was to compare the change in trunk fat mass (g) between insulin detemir versus insulin NPH at baseline and at week 26. A standard deviation of 5% was chosen based on a previous trial. A difference in trunk fat mass of 5% was considered clinically relevant also according to this trial; Test type: Superiority or Other; p = 0.849, ANCOVA — H01 (hypothesis): Micro detemir = micro NPH against the alternative H01: Microl detemir ≠ micro NPH; Mean Difference (Final Values) = -0.645, 95% CI [-7.404 to 6.114], Standard Error of Mean 3.364

2. Primary Outcome: Percentage Change in Trunk Fat Mass (Defined as Peripheral Fat Ratio)
Description: as for outcome 1
Time Frame: week 0, week 26
Population: Per protocol (PP) population: All randomised and exposed subjects who completed the 26-week treatment without significantly deviating from the inclusion/exclusion criteria and the withdrawal criteria or other aspects of the protocol considered to potentially affect the efficacy results. Compared to the ITT population, two subjects were excluded.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 21 | 31
percent change | 0.535 (2.875) | 1.126 (2.212)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.948, ANCOVA — H01: Micro detemir = micro NPH against the alternative H01: Microl detemir ≠ micro NPH; Mean Difference (Final Values) = -0.590, 95% CI [-7.588 to 6.407], Standard Error of Mean 3.478

3. Primary Outcome: Absolute Change in Trunk Fat Mass
Description: Absolute change in trunk fat mass as response variable with treatment, sex and Metformin use as fixed factors, and trunk fat mass at week 0 as covariate.
Time Frame: week 0, week 26
Population: ITT analysis set using LOCF is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in the change in trunk fat mass at week 26.
Measure: Least Squares Mean (Standard Error); unit: grams (g)
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
grams (g) | 133.99 (412.88) | -62.37 (320.00)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.696, ANCOVA — H01: Micro detemir = micro NPH against the alternative H01: Microl detemir ≠ micro NPH; Mean Difference (Final Values) = 196.36, 95% CI [-805.8 to 1198.5], Standard Error of Mean 498.70

4. Primary Outcome: Absolute Change in Trunk Fat Mass
Description: as for outcome 3
Time Frame: week 0, week 26
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: grams (g)
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 21 | 31
grams (g) | 153.38 (423.93) | 39.43 (327.78)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.710, ANCOVA — H01: Micro detemir = micro NPH against the alternative H01: Microl detemir ≠ micro NPH; Mean Difference (Final Values) = 192.81, 95% CI [-844.0 to 1229.7], Standard Error of Mean 515.40

5. Secondary Outcome: Absolute Change in Whole Body Fat Mass
Description: Absolute change in whole body fat mass as response variable with treatment, sex and Metformin use as fixed factors, and trunk fat mass at week 0 as covariate.
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in the change in whole body fat mass at week 26.
Measure: Least Squares Mean (Standard Error); unit: grams (g)
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
grams (g) | 1147.1 (635.79) | 858.88 (494.14)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.709, ANCOVA; Mean Difference (Final Values) = 288.21, 95% CI [-1252.0 to 1828.4], Standard Error of Mean 766.41

6. Secondary Outcome: Percentage Change in Whole Body Fat Mass
Description: Percentage Change in Whole Body Fat Mass as response variable with treatment, sex and Metformin use as fixed factors, and whole Body Fat Mass at week 0 as covariate.
Time Frame: Week 0, week 26
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
percent change | 3.870 (2.267) | 4.047 (1.762)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.948, ANCOVA; Mean Difference (Final Values) = -0.178, 95% CI [-5.668 to 5.313], Standard Error of Mean 2.732

7. Secondary Outcome: Absolute Change in Whole Body Lean Mass
Description: Absolute change in whole body lean mass as response variable with treatment, sex and Metformin use as fixed factors, whole body lean mass at week 0 as covariate.
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in the change in whole body lean mass at week 26.
Measure: Least Squares Mean (Standard Error); unit: grams (g)
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
grams (g) | -54.20 (673.32) | 1097.2 (524.74)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.162, ANCOVA; Mean Difference (Final Values) = -1151.0, 95% CI [-2780.0 to 477.33], Standard Error of Mean 810.48

8. Secondary Outcome: Percentage Change in Whole Body Lean Mass
Description: Percentage Change in Whole Body Lean Mass as response variable with treatment, sex and Metformin use as fixed factors, and whole Body Lean Mass at week 0 as covariate.
Time Frame: Week 0, week 26
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
percent change | 0.051 (1.485) | 2.798 (1.158)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.131, ANCOVA; Mean Difference (Final Values) = -2.747, 95% CI [-6.340 to 0.846], Standard Error of Mean 1.788

9. Secondary Outcome: Absolute Change in Trunk Lean Mass
Description: Absolute change in trunk lean mass as response variable with treatment, sex and Metformin use as fixed factors, and trunk lean mass at week 0 as covariate
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in the change in trunk lean mass at week 26.
Measure: Least Squares Mean (Standard Error); unit: grams (g)
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
grams (g) | 359.43 (306.47) | 469.84 (238.67)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.766, ANCOVA; Mean Difference (Final Values) = -110.4, 95% CI [-851.3 to 630.51], Standard Error of Mean 368.69

10. Secondary Outcome: Percentage Change in Trunk Lean Mass
Description: Percentage Change in Trunk Lean Mass as response variable with treatment, sex and Metformin use as fixed factors, and Trunk Lean Mass at week 0 as covariate.
Time Frame: Week 0, week 26
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
percent change | 1.480 (1.381) | 2.090 (1.076)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.716, ANCOVA; Mean Difference (Final Values) = -0.610, 95% CI [-3.949 to 2.729], Standard Error of Mean 1.662

11. Secondary Outcome: Absolute Change in Calculated Whole Body Fat Percentage
Description: Absolute change in calculated whole body fat percentage as response variable with treatment, sex and Metformin use as fixed factors, and calculated whole body fat percentage at week 0 as covariate
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in the calculated whole body fat percentage at week 26.
Measure: Least Squares Mean (Standard Error); unit: percent of whole body fat (%)
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
percent of whole body fat (%) | 0.782 (0.578) | 0.291 (0.450)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.483, ANCOVA; Mean Difference (Final Values) = 0.491, 95% CI [-0.906 to 1.888], Standard Error of Mean 0.695

12. Secondary Outcome: Percentual Change in Calculated Whole Body Fat Percentage
Description: Percentual Change in Calculated Whole Body Fat Percentage as response variable with treatment, sex and Metformin use as fixed factors, and Calculated Whole Body Fat Percentage at week 0 as covariate.
Time Frame: Week 0, week 26
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
percent change | 1.607 (1.587) | 1.491 (1.235)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.952, ANCOVA; Mean Difference (Final Values) = 0.116, 95% CI [-3.721 to 3.953], Standard Error of Mean 1.909

13. Secondary Outcome: Absolute Change in Calculated Trunk Fat Percentage
Description: Absolute change in calculated trunk fat percentage as response variable with treatment, sex and Metformin use as fixed factors, and calculated trunk fat percentage at week 0 as covariate
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in the calculated trunk fat percentage at week 26.
Measure: Least Squares Mean (Standard Error); unit: percent of trunk fat (%)
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
percent of trunk fat (%) | -0.600 (0.621) | -0.321 (0.483)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.711, ANCOVA; Mean Difference (Final Values) = -0.278, 95% CI [-1.778 to 1.221], Standard Error of Mean 0.746

14. Secondary Outcome: Percentual Change in Calculated Trunk Fat Percentage
Description: Percentual Change in Calculated Trunk Fat Percentage as response variable with treatment, sex and Metformin use as fixed factors, and Calculated Trunk Fat Percentage at week 0 as covariate.
Time Frame: Week 0, week 26
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
percent change | -1.543 (1.542) | 0.042 (1.201)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.397, ANCOVA; Mean Difference (Final Values) = -1.585, 95% CI [-5.310 to 2.141], Standard Error of Mean 1.854

15. Secondary Outcome: Absolute Change in Visceral Adipose Tissue Area
Description: Absolute change in visceral adipose tissue area as response variable with treatment, sex and Metformin use as fixed factors, and visceral adipose tissue area at week 0 as covariate
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in the visceral adipose tissue area at week 26.
Measure: Least Squares Mean (Standard Error); unit: cm^2
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
cm^2 | -3.258 (9.122) | 5.658 (7.042)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.421, ANCOVA; Mean Difference (Final Values) = -8.916, 95% CI [-30.99 to 13.159], Standard Error of Mean 10.985

16. Secondary Outcome: Percentage Change in Visceral Adipose Tissue Area
Description: Percentage Change in Visceral Adipose Tissue Area as response variable with treatment, sex and Metformin use as fixed factors, and Visceral Adipose Tissue Area at week 0 as covariate.
Time Frame: Week 0, week 26
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
percent change | -0.535 (5.162) | 4.526 (3.4985)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.420, ANCOVA; Mean Difference (Final Values) = -5.061, 95% CI [-17.55 to 7.430], Standard Error of Mean 6.216

17. Secondary Outcome: Absolute Change in Subcutaneous Adipose Tissue Area
Description: Absolute change in subcutaneous adipose tissue area as response variable with treatment, sex and Metformin use as fixed factors, and subcutaneous adipose tissue area at week 0 as covariate
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in the subcutaneous adipose tissue area at week 26.
Measure: Least Squares Mean (Standard Error); unit: cm^2
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
cm^2 | 7.654 (10.764) | 12.616 (8.375)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.705, ANCOVA; Mean Difference (Final Values) = -4.961, 95% CI [-31.10 to 21.178], Standard Error of Mean 13.007

18. Secondary Outcome: Percentage Change in Subcutaneous Adipose Tissue Area
Description: Percentage Change in Subcutaneous Adipose Tissue Area as response variable with treatment, sex and Metformin use as fixed factors, and Subcutaneous Adipose Tissue Area at week 0 as covariate.
Time Frame: Week 0, week 26
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
percent change | 1.153 (3.952) | 5.743 (3.075)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.341, ANCOVA; Mean Difference (Final Values) = -4.590, 95% CI [-14.19 to 5.007], Standard Error of Mean 4.776

19. Secondary Outcome: Absolute Change in Calculated Visceral/Subcutaneous Adipose Tissue Ratio
Description: Absolute change in Calculated Visceral/Subcutaneous Adipose Tissue Ratio as response variable with treatment, sex and Metformin use as fixed factors, and Calculated Visceral/Subcutaneous Adipose Tissue Area at week 0 as covariate.
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in the calculated Visceral /Subcutaneous adipose tissue ratio at week 26.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
ratio | -0.032 (0.028) | -0.036 (0.022)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.902, ANCOVA; Mean Difference (Final Values) = 0.004, 95% CI [-0.064 to 0.073], Standard Error of Mean 0.034

20. Secondary Outcome: Percentage Change in Calculated Visceral/Subcutaneous Adipose Tissue Ratio
Description: Percentage Change in Calculated Visceral/Subcutaneous Adipose Tissue Area as response variable with treatment, sex and Metformin use as fixed factors, and Calculated Visceral/Subcutaneous Adipose Tissue Area at week 0 as covariate.
Time Frame: Week 0, week 26
Population: as for outcome 19
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
percent change | -4.092 (3.211) | -3.303 (2.493)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.839, ANCOVA; Mean Difference (Final Values) = -0.789, 95% CI [-8.525 to 6.947], Standard Error of Mean 3.850

21. Secondary Outcome: Absolute Change in Liver/Spleen Attenuation Ratio
Description: Absolute change in Liver/Spleen Attenuation Ratio as response variable with treatment, sex and Metformin use as fixed factors, and Liver/Spleen Attenuation Ratio at week 0 as covariate.
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and four subjects in the Insulin NPH group did not present a value in the liver to spleen attenuation ratio at week 26.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 31
ratio | -0.044 (0.035) | -0.023 (0.026)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.607, ANCOVA; Mean Difference (Final Values) = -0.021, 95% CI [-0.105 to 0.062], Standard Error of Mean 0.041

22. Secondary Outcome: Percentage Change in Liver/Spleen Attenuation Ratio
Description: Percentage Change in Liver/Spleen Attenuation Ratio as response variable with treatment, sex and Metformin use as fixed factors, and Liver to Spleen Attenuation Ratio at week 0 as covariate.
Time Frame: Week 0, week 26
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 31
percent change | -2.632 (3.102) | -0.855 (2.355)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.635, ANCOVA; Mean Difference (Final Values) = -1.777, 95% CI [-9.254 to 5.700], Standard Error of Mean 3.719

23. Secondary Outcome: Absolute Change in HbA1c (Glycosylated Haemoglobin)
Description: Absolute Change in HbA1c as response variable with treatment, sex and Metformin use as fixed factors, and HbA1c at week 0 as covariate.
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set using LOCF (Last Observation Carried Forward) is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in the hbA1c at week 26.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
percentage of glycosylated haemoglobin | -0.922 (0.226) | -0.792 (0.172)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.628, ANCOVA; Mean Difference (Final Values) = -0.130, 95% CI [-0.663 to 0.403], Standard Error of Mean 0.266

24. Secondary Outcome: Absolute Change in Fasting Plasma Glucose (FPG)
Description: Absolute Change in Fasting Plasma Glucose as response variable with treatment, sex and Metformin use as fixed factors, and Fasting Plasma Glucose at week 0 as covariate.
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set using LOCF (Last Observation Carried Forward) is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and six subjects in the Insulin NPH group did not present a value in the fasting plasma glucose at week 26.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 29
mg/dL | -48.29 (14.599) | -37.36 (11.616)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.535, ANCOVA; Mean Difference (Final Values) = -10.92, 95% CI [-46.03 to 24.182], Standard Error of Mean 17.460

25. Secondary Outcome: Absolute Change in Adiponectin
Description: Absolute change in adiponectin as response variable with treatment, sex and Metformin use as fixed factors, and Adiponectic at week 0 as covariate.
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Six subjects in the Insulin Detemir group and four subjects in the Insulin NPH group did not present a value in the adiponectin at week 26.
Measure: Least Squares Mean (Standard Error); unit: mcg/dL
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 18 | 31
mcg/dL | 0.926 (3.605) | 2.844 (2.641)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.660, ANCOVA; Mean Difference (Final Values) = -1.918, 95% CI [-10.65 to 6.813], Standard Error of Mean 4.332

26. Secondary Outcome: Absolute Change in Total Cholesterol
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Three subjects in the Insulin Detemir group and four subjects in the Insulin NPH group did not present a value in the total cholesterol at week 26.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 21 | 31
mg/dL | -8.96 (57.60) | 7.77 (31.47)

27. Secondary Outcome: Absolute Change in High Density Lipoprotein (HDL) Cholesterol
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Three subjects in the Insulin Detemir group and four subjects in the Insulin NPH group did not present a value in the HDL cholesterol at week 26.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 21 | 31
mg/dL | -0.95 (7.94) | 2.87 (7.46)

28. Secondary Outcome: Absolute Change in Low Density Lipoprotein (LDL) Cholesterol
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Three subjects in the Insulin Detemir group and four subjects in the Insulin NPH group did not present a value in the LDL cholesterol at week 26.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 21 | 31
mg/dL | 2.39 (24.63) | 6.14 (26.74)

29. Secondary Outcome: Absolute Change in Very Low Density Lipoprotein (VLDL) Cholesterol
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Three patients in the Insulin Detemir group and seven patients in the Insulin NPH group did not present a value in the VLDL cholesterol at week 26.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 21 | 28
mg/dL | 1.05 (12.08) | 1.54 (10.29)

30. Secondary Outcome: Absolute Change in Triglycerides
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Three patients in the Insulin Detemir group and six patients in the Insulin NPH group did not present a value in the triglycerides at week 26.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 21 | 29
mg/dL | -14.71 (57.60) | -20.97 (70.73)

31. Secondary Outcome: Absolute Change in Free Fatty Acids
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and four subjects in the Insulin NPH group did not present a value in the free fatty acids at week 26.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 31
mg/dL | -0.03 (0.20) | -0.05 (6.01)

32. Secondary Outcome: Absolute Change in Haemoglobin
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and four subjects in the Insulin NPH group did not present a value in the haemoglobin at week 26.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 31
g/dL | -0.38 (0.75) | -0.35 (0.86)

33. Secondary Outcome: Absolute Change in Blood Volume (Haematocrit)
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and four subjects in the Insulin NPH group did not present a value in the Haematocrit at week 26.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 31
percentage | -1.17 (2.49) | -1.06 (2.24)

34. Secondary Outcome: Absolute Change in Thrombocytes
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Only one subjects in the Insulin Detemir group presented values at week 26 in thrombocytes, whilst no subjects showed available values at week 26 in the Insulin NPH group.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 1 | 0
percentage | 0.10 (NA) — No standard deviation calculated due to lack of available values at week 26 |

35. Secondary Outcome: Absolute Change in Erythrocytes
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and four subjects in the Insulin NPH group did not present a value in Erythrocytes at week 26.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 21 | 31
percentage | 4.64 (0.58) | 4.38 (0.43)

36. Secondary Outcome: Absolute Change in Leucocytes
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and four subjects in the Insulin NPH group did not present a value in Leucocytes at week 26.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 31
10^9 cells/L | -0.01 (1.68) | -0.07 (1.17)

37. Secondary Outcome: Absolute Change in Lymphocytes
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Only one subject in the Insulin Detemir group presented values at week 26 in Lymphocytes, whilst no subjects showed available values at week 26 in the Insulin NPH group.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 1 | 0
percentage | -0.10 (NA) — No standard deviation calculated due to lack of available values at week 26 |

38. Secondary Outcome: Absolute Change in Monocytes
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Only one subject in the Insulin Detemir group presented values at week 26 in Monocytes, whilst no subjects showed available values at week 26 in the Insulin NPH group.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 1 | 0
percentage | 0.10 (NA) — No standard deviation calculated due to lack of available values at week 26 |

39. Secondary Outcome: Absolute Change in Neutrophils
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. The comparison between visits could only be done with nine subjects in the Insulin Detemir group since only these patients had values available at week 0 and at week 26 while this applied to 22 subjects in the Insulin NPH group.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 9 | 22
percentage | -0.29 (1.32) | 0.01 (1.03)

40. Secondary Outcome: Absolute Change in Eosinophils
Time Frame: Week 0, week 26
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 9 | 22
10^9 cells/L | 0.01 (0.08) | 0.01 (0.09)

41. Secondary Outcome: Absolute Change in Basophils
Time Frame: Week 0, week 26
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 9 | 22
10^9 cells/L | 0.00 (0.10) | -0.01 (0.05)

42. Secondary Outcome: Absolute Change in Creatinine
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in the Creatinine at week 26.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
mg/dL | 0.03 (0.19) | -0.00 (0.16)

43. Secondary Outcome: Absolute Change in Creatine Phosphokinase
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in the Creatine Phosphokinase at week 26.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
IU/L | -19.86 (71.49) | 21.56 (50.11)

44. Secondary Outcome: Absolute Change in Urea
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in the Urea at week 26.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
mg/dL | 2.45 (10.00) | 0.50 (6.75)

45. Secondary Outcome: Absolute Change in Albumin
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group did not present an albumin baseline value and another two at week 26 and four subjects in the Insulin NPH group did not present a value in the albumin at week 26.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 20 | 31
mg/dL | -0.02 (0.40) | 0.01 (0.37)

46. Secondary Outcome: Absolute Change in Bilirubin Total
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in the Bilirubin Total at week 26.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
mg/dL | -0.07 (0.23) | -0.07 (0.20)

47. Secondary Outcome: Absolute Change in Alanine Aminotransferase (ALAT)
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and four subjects in the Insulin NPH group did not present a value in the ALAT at week 26.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 31
IU/L | -3.59 (8.43) | -4.55 (19.68)

48. Secondary Outcome: Absolute Change in Aspartate Aminotransferase (ASAT)
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and four subjects in the Insulin NPH group did not present a value in the ASAT at week 26.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 31
IU/L | 0.23 (6.91) | -0.48 (12.87)

49. Secondary Outcome: Absolute Change in Alkaline Phosphatase
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. One subject in the Insulin Detemir group did not present an albumin baseline value and another two at week 26 and four subjects in the Insulin NPH group did not present a value in the Alkaline Phosphatase at week 26.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 21 | 31
IU/L | -7.10 (18.61) | -12.55 (57.55)

50. Secondary Outcome: Absolute Change in Sodium
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Two subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in Sodium at week 26.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 32
mmol/L | 1.12 (3.81) | 0.69 (6.02)

51. Secondary Outcome: Absolute Change in Potassium
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Three subjects in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in Potassium at week 26.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 21 | 32
mmol/L | -0.20 (0.97) | 0.21 (0.83)

52. Secondary Outcome: Absolute Change in Body Weight
Description: Absolute change in body weight was based on ANCOVA model for absolute change from week 0 to week 26 as response variable with treatment, sex and Metformin use as fixed factors, and body weight at week 0 as covariable.
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. One subject in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in body weight at week 26.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 23 | 32
kg | 1.663 (0.779) | 2.293 (0.630)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.518, ANCOVA; Mean Difference (Final Values) = -0.629, 95% CI [-2.572 to 1.313], Standard Error of Mean 0.967

53. Secondary Outcome: Absolute Change in Waist Circumference
Description: Absolute change in waist circumference was based on ANCOVA model for absolute change from week 0 to week 26 as response variable with treatment, sex and Metformin use as fixed factors, and Waist at week 0 as covariate.
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. One subject in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in waist circumference at week 26.
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 23 | 32
cm | 0.064 (1.062) | 0.609 (0.832)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.673, ANCOVA; Mean Difference (Final Values) = -0.546, 95% CI [-3.123 to 2.032], Standard Error of Mean 1.283

54. Secondary Outcome: Absolute Change in Hip Circumference
Description: Absolute Change in Hip Circumferences was based on ANCOVA model for absolute change from week 0 to week 26 as response variable with treatment, sex, and Metformin use as fixed factors, and hip circumference at week 0 as covariate.
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. One subject in the Insulin Detemir group and three subjects in the Insulin NPH group did not present a value in hip circumference at week 26.
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 23 | 32
cm | 0.577 (1.142) | 0.112 (0.905)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.738, ANCOVA; Mean Difference (Final Values) = 0.466, 95% CI [-2.319 to 3.250], Standard Error of Mean 1.386

55. Secondary Outcome: Absolute Change in hsCRP (Highly Sensitive C Reactive Protein)
Description: Absolute change in hsCRP was based on ANCOVA model for absolute change from week 0 to week 26 as response variable with treatment, sex and Metformin use as fixed factors, and hsCRP at week 0 as covariate.
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. One subject from each treatment group did not present a hsCRP available value at week 0. Two subjects from the Insulin Detemir group and three subjects from the Insulin NPH group did not show a hsCRP available value at week 26.
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 21 | 31
mg/L | 1.200 (1.787) | -0.862 (1.373)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.346, ANCOVA; Mean Difference (Final Values) = 2.062, 95% CI [-2.300 to 6.423], Standard Error of Mean 2.168

56. Secondary Outcome: Absolute Change in PAI-1 (Plasminogen Activator Inhibitor-1)
Time Frame: Week 0, week 26
Population: Intention-To-Treat (ITT) analysis set is all randomised subjects exposed to at least one dose of the trial product. Three subjects from the Insulin Detemir group and one subject from the Insulin NPH group did not show a PAI-1 available value at week 0. Three subjects from each treatment group did not present a PAI-1 available value at week 26.
Measure: Least Squares Mean (Standard Error); unit: ng/L
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 18 | 31
ng/L | -10.77 (5.119) | -12.50 (3.765)
Statistical Analysis 1: Comparison: Insulin Detemir vs Insulin NPH; Test type: Superiority or Other; p = 0.781, ANCOVA; Mean Difference (Final Values) = 1.726, 95% CI [-10.71 to 14.167], Standard Error of Mean 6.173

57. Secondary Outcome: Number of Hypoglycaemic Episodes
Description: Number of episodes reported during the trial.
Time Frame: Weeks 0-26
Population: Full analysis set is all randomised subjects who were exposed at least one dose of the trial product.
Measure: Number; unit: episodes
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 24 | 35
episodes | 17 | 32

58. Secondary Outcome: Number of Non-serious Adverse Events
Description: Number of episodes reported during the trial.
Time Frame: Weeks 0-26
Population: Full analysis set is all randomised subjects who were exposed at least one dose of the trial product.
Measure: Number; unit: events
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 24 | 35
events | 64 | 103

ADVERSE EVENTS:
Time Frame: Adverse events were collected in a time span of 26 weeks.
Description: Safety analysis set is all randomised subjects exposed to at least one dose of trial drug(s).
Arm/Group | Insulin Detemir | Insulin NPH
Serious Adverse Events (participants affected / at risk) | 3/24 | 3/35
Other Adverse Events (participants affected / at risk) | 18/24 | 29/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (N=24) | Insulin NPH (N=35)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insulin aspart overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Crushed vertebra D-12 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
White carotid ictus (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic cardiopathy (Cardiac disorders) | 1 (1) | 0 (0)
Vascular ulcer worsening (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (N=24) | Insulin NPH (N=35)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Abdominal pain, upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Pain (General disorders) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 3 (4)
Ear infection (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 7 (11) | 7 (9)
Pharyngitis (Infections and infestations) | 0 (0) | 3 (3)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (10)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 7 (7)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other